







## **CONSENT FORM** (Final version 1.1: 25 March 2020)

Title of Study: Molecular Pathways Involved in Knee Pain

**IRAS Project ID: 275727** 

Name of Chief Investigator: Doctor Ana Valdes, Associate Professor and Reader

Name of Participant:

| | | Pleas | se initia | l box |
|---|---|---|---|---|
| 1. | . I confirm that I have read and understand the information sheet version number x.x xx/xx/xxxx for the above study. I have had the opportunity to consider the informatio questions and have had these answered satisfactorily. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, v giving any reason, and without my medical care or legal rights being affected. I understar should I withdraw, then the information collected so far cannot be erased and the information may still be used in the project analysis. | nd that | | |
| 3. | I understand that relevant sections of my medical notes and data collected in the study noted at by authorised individuals from the University of Nottingham, the research groundly and regulatory authorities where it is relevant to my taking part in this study, permission for these individuals to have access to these records and to collect, store, and publish information obtained from my participation in this study. I understand the personal details will be kept confidential. | up, the<br>I give<br>nalyse | | |
| 4. | . I understand that synovial fluid will be taken from my knee joint. | | | |
| 5. | I agree that the samples I have given and the information gathered about me can be sto the University of Nottingham for possible use in future studies. I understand that my sa could be involved in the analysis and use of human DNA and may be shared with other conduct medical research such as universities, research institutes or pharmac companies. Any samples or data used will be anonymised, and I will not be identified way. [OPTIONAL] | amples<br>centres<br>eutical | YES | NO NO |
| 6. | . I agree to undertake the extra clinical assessment and take part in the sub-study. [OPTIC | )NAL] | | |
| 7. | ี้. I agree to be further contacted in the future to be informed about this or new research. [opา | ΓΙΟΝΑL] | YES | NO |
| 8. | . I agree to take part in the above study. | | | |
| <br>Na | lame of Participant Date Signature | | | |
| <del></del> | Determine the second se | | | |
| 1NS | lame of Person taking consent Date Signature | | | |